CLINICAL TRIAL: NCT03872336
Title: Acute Labetalol Use in Preeclampsia Randomized Trial
Brief Title: Acute Labetalol Use in Preeclampsia
Acronym: ALERT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5254
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Preeclampsia With Severe Features
Keywords: Hypertension; Labetalol; Obesity
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principle investigator and outcomes assessor are masked to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental labetalol dose (Experimental): Subjects receive 40mg, 60mg 80mg in succession after each severe BP
  Interventions: Drug: Experimental labetalol dose
- Current standard of care (Active Comparator): Subjects receive 20mg, 40mg 80mg in succession after each severe BP
  Interventions: Other: Current standard of care

INTERVENTIONS:
Drug: Experimental labetalol dose — Subjects who have sustained severe hypertension (SBP≥160 mmHg and/or DBP≥110 mmHg), 15 min apart receive the experimental dosing of labetolol. Subjects in both groups are managed following the standard guidelines established by ACOG (Committee Opinion #623). For each successive episode of hypertension treatment, patients are asked a set of questions to monitor for adverse medication side-effects. The fetus is electronically monitored for four hours after the last IV dose.
  Arms: Experimental labetalol dose
Other: Current standard of care — Subjects who have sustained severe hypertension (SBP≥160 mmHg and/or DBP≥110 mmHg), 15 min apart receive the standard dosing of labetolol. Subjects in both groups are managed following the standard guidelines established by ACOG (Committee Opinion #623). For each successive episode of hypertension treatment, patients are asked a set of questions to monitor for adverse medication side-effects. The fetus is electronically monitored for four hours after the last IV dose.
  Arms: Current standard of care

SUMMARY:
The purpose of this study is to understand if administration of a personalized dose of the anti-hypertensive medication, labetalol, based on patient's body-mass index, will be more effective at controlling severe hypertension during pregnancy, compared to the current standard dosing.

DETAILED DESCRIPTION:
The investigators seek to asses the effect of obesity (BMI>30) on severe hypertension control in patients with preeclampsia with severe features. The investigators hypothesize that successive administration of 40-60-80 mg of labetolol will reduce time to blood pressure control versus the standard dosing, 20-40-80 mg labetolol, recommended by the American College of Obstetricians and Gynecologists in 2015.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30
* Age ≥ 18 years
* Gestational age ≥ 24 weeks
* Singleton gestation
* One sustained severe range blood pressure at Albany Medical Center

Exclusion Criteria:

* Known allergic reaction to labetlol
* Persistent mild-moderate asthma (≥ 2 rescue inhaler uses per week in the previous month)
* Obstructive airway disease
* Bradycardia < 70 beats/min
* Heart block > 1st degree or history of heart failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Time to blood pressure control | 4 hours after last labetalol dosing
  The length of time the subject continued to have non-severe range blood pressure following administration of labetolol.

SECONDARY OUTCOMES:
Differences in racial response | 4 hours after last labetalol dosing
  The difference in time for blood pressure control amongst racial groups
Maternal adverse events | within 3 months of delivery
  Anticipated and unanticipated maternal events including Symptomatic hypotension, bradsycardia, bronchospam, seizure, stroke, death
Neonatal adverse events | within 28 days of delivery
  complications experienced by the neonate including PGAR score < 5, need for respiratory support, blood glucose, death

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Obstetrics and Gynecology, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Committee Opinion No. 623: Emergent therapy for acute-onset, severe hypertension during pregnancy and the postpartum period. Obstet Gynecol. 2015 Feb;125(2):521-525. doi: 10.1097/01.AOG.0000460762.59152.d7. PMID 25611642